CLINICAL TRIAL: NCT02710058
Title: Experience of Arab American Women With Breast Cancer: In-depth Interviews A Qualitative Study to Explore the Influence of the Arab Culture on Coping With Breast Cancer
Brief Title: Experience of Arab American Women With Breast Cancer: In-depth Interviews
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-246
Record Dates: First submitted 2016-03-03; First posted 2016-03-16 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: support group; 15-246; The Arab American Breast Cancer Education and Referral Program (AMBER)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Arab American Women with Breast Cancer: We conducted a study using an evaluation assessment survey to assess the impact of the AMBER support groups on quality of life parameters, compliance with treatment appointments, and patient/family support. After reviewing preliminary results, we identified several recurrent themes, such as the need for health information, discrepancies around the extent of family support and disease disclosure, and an overall satisfaction with the support groups. To further examine these themes, we are initiating a qualitative research study using an in-depth interview guide. A trained interviewer bilingual in Arabic and English will conduct 10-15 in-depth interviews, to saturation, with AMBER's support group participants over a 6 month period.
  Interventions: Behavioral: one-time qualitative assessment

INTERVENTIONS:
Behavioral: one-time qualitative assessment — The study involves a one-time qualitative assessment to explore key cultural influences on AMBER breast cancer survivors' health behavior. We will focus on self-efficacy in healthcare, coping with breast cancer, social networks of support, and culturally-sensitive support groups. The study investigator will administer questions from the structured interview guide, estimated to take 90 minutes.

SUMMARY:
The investigators are conducting a study entitled 'Experience of Arab American Women with Breast Cancer: In-depth Interviews' through which they hope to learn more about Arab women's experience with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* AMBER participant diagnosed with breast cancer who attended at least 1 support group meeting
* Aged 18 to 85
* Arabic-speaking

Exclusion Criteria:

None

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is open to current and previous AMBER support group participants held at the MSK Brooklyn Infusion Center.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Understanding the influence of Arab culture on health behavior | 6 months
  particularly with regard to breast cancer by in-depth interviews

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gany, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- MSKCC Brooklyn Infusion Center, Brooklyn, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/